CLINICAL TRIAL: NCT05223400
Title: Drug Use Evaluation Study of Clindamycin in Critical Care Units in Alexandria Main University Hospital
Brief Title: Drug Use Evaluation of Clindamycin in Critical Care Units in Alexandria Main University Hospital
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Heba Shaker, supervisor of clinical pharmacy unit in Alexandria Main University Hospital, Alexandria University
Other Study IDs: 0305292
Record Dates: First submitted 2022-01-06; First posted 2022-02-04 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Infection, Bacterial
MeSH Terms: conditions — Bacterial Infections | interventions — Clindamycin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Clindamycin Injection — it is a clindamycin use evaluation study

SUMMARY:
Irrational use of antibiotics is a one of the main health system problems,it leads to antibiotic resistance,increasing antibiotics side effects and the total cost. This study is a medication use evaluation study aims to evaluate intravenous clindamycin prescribing practice in critical care units in Alexandria Main University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years old or more .
* Patients on clindamycin as an empirical treatment.
* Patients started clindamycin as an emperical treatment in other departments but the physician approved to continue it in critical care.

Exclusion Criteria:

* Children (less than 18 years old)
* Patients started clindamycin as a defenitive treatment (based on microbiological culture results).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to critical care units and on clindamycin emperical therapy .
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
the number of prescriptions with appropriate indications of clindamycin will be counted during the retrospective observation of all prescriptions | 1 month
  appropriateness of clindamycin indication will be determined according to IDSA guidelines.

SECONDARY OUTCOMES:
the number of prescriptions with duplication of therapy with clindamycin will be counted during the retrospective observation of all prescriptions | 1 month
  duplication of therapy means prescribing of clindamycin concurrently with another antibiotic to target the same microorganism.
the number of patients who had diarrhea as a main side effect of clindamycin | 1 month
  diarrhea is a main side effect of clindamycin so in the study the number of patients who had diarrhea will be counted during the retrospective observation of all prescriptions
the number of patients who had severe drug interactions with clindamycin | 1 month
  in the study the number of patients who severe clindamycin drugs interactions will be counted during the retrospective observation of all prescriptions
Total clindamycin DDD defined daily doses and clindamycin defined daily doses per 1000 patients days. | 1 month
  Defined daily doses measurement of a drug is an indicator put by WHO , it indicates the consumption of this drug in a hospital or a department and defined daily doses per 1000 patients days indicates the consumption of this drug in relation to the total number of patients in a certain period of time.
to calculate the total cost of clindamycin. | 1 month
  The cost of clindamycin treatment courses of all patients will be calculated in the Egyptian pound

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Mdicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes